CLINICAL TRIAL: NCT02193035
Title: Microparticles as an Inflammatory Marker in Severe Aortic Stenosis.
Brief Title: Microparticles in Severe Aortic Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Pedro A. Lemos, Professor of Medicine, InCor Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 31446114.1.0000.0068
Record Dates: First submitted 2014-07-11; First posted 2014-07-17 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Aortic Valve Stenosis
Keywords: Microparticles; Severe aortic stenosis; Calcified aortic stenosis; transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group (Experimental): Patients with severe aortic stenosis treated with transcatheter aortic valve replacement (TAVR). Microparticle levels will be measured before and after TAVR.
  Interventions: Other: Microparticle levels

INTERVENTIONS:
Other: Microparticle levels — Microparticle levels will be evaluated with flow cytometry and nanoparticle tracking analysis

SUMMARY:
Microparticles are small cell fragments that can induce fat plaques, calcification and formation of thrombus. They can be released through multiple stimulations, but also the high flow of blood through partially obstructed aortic valves.

In patients with severely obstructed aortic valves the investigators hypothesize that microparticles levels will be elevated and that they will go down after percutaneous treatment of the valves.

DETAILED DESCRIPTION:
Microparticle (MPs) levels and subtypes according to endothelial cell, macrophage and platelet markers will be measured by flow-cytometry using appropriate fluorochromes. Patient baseline (including measures of severity of aortic stenosis and its calcification), procedural data, and clinical evolution will be collected. Inflammatory markers will be measured, which along with clinical date will be tested for correlation with microparticle levels.

Patients MPs will be measured before and after percutaneous treatment of the severe aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication to be treated with transcatheter aortic valve replacement.

Exclusion Criteria:

* Non native aortic valve
* Moderate aortic regurgitation
* The following complications following valve implantation: patient instability, need for vasoactive pressors, sepsis and severe infections, stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Difference in microparticle levels | Day 5
  Difference of total microparticle levels before and after treatment of patients with percutaneous aortic valve replacement

SECONDARY OUTCOMES:
Endothelial microparticle levels | Day 5
  Difference of endothelial microparticle levels before and after treatment of patients with percutaneous aortic valve replacement
Macrophage microparticle levels | Day 5
  Difference of macrophage microparticle levels before and after treatment of patients with percutaneous aortic valve replacement
Platelet microparticle levels | Day 5
  Difference of platelet microparticle levels before and after treatment of patients with percutaneous aortic valve replacement

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Lemos, MD PhD, Study Chair — Heart Institute - InCor. University of Sao Paulo Medical School; Julio F Marchini, MD PhD, Principal Investigator — Heart Institute - InCor. University of Sao Paulo Medical School
Locations (1):
- Heart Institute - InCor. University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marchini JF, Miyakawa AA, Tarasoutchi F, Krieger JE, Lemos P, Croce K. Endothelial, platelet, and macrophage microparticle levels do not change acutely following transcatheter aortic valve replacement. J Negat Results Biomed. 2016 Apr 11;15:7. doi: 10.1186/s12952-016-0051-2. PMID 27063005